CLINICAL TRIAL: NCT06997692
Title: Effect of Gongs Mobilization With Neuromuscular Electrical Stimulation vs Conservative Exercises Among Adhesive Capsulitis
Brief Title: Effect of Gongs Mobilization With Neuromuscular Electrical Stimulation vs Conservative Exercises Among AC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/823
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's Mobilization with NMES (Experimental)
  Interventions: Diagnostic Test: Gong's Mobilization with NMES
- Comprehensive Conservative Physical Therapy (Active Comparator)
  Interventions: Combination Product: Comprehensive Conservative Physical Therapy

INTERVENTIONS:
Diagnostic Test: Gong's Mobilization with NMES — Gong's Mobilization Technique: The participant will be positioned in a side-lying posture on a height-adjustable bed, with the affected side upward and the head supported by a pillow The therapist will apply an antero-posterior glide to the humeral head while stabilizing the scapula with the other hand. The participant will perform quick, powerful shoulder abduction in the coronal plane without external rotation or elbow flexion while the therapist maintains the mobilization force.
  Arms: Gong's Mobilization with NMES
Combination Product: Comprehensive Conservative Physical Therapy — Thermal Modality Application: Participants will receive either a cold or hot pack (based on individual preference and clinical presentation) applied to the affected shoulder for 10-15 minutes. Cold packs will be wrapped in a thin towel and applied to
  Arms: Comprehensive Conservative Physical Therapy

SUMMARY:
This study evaluates the effectiveness of Gong's mobilization combined with neuromuscular electrical stimulation versus conservative exercises in improving range of motion, pain relief, and functional outcomes in patients with adhesive capsulitis.

DETAILED DESCRIPTION:
Using a randomized controlled design with 36 participants with estimated drop out 10% will be 40, the study will measure changes in active and passive shoulder mobility and SPADI scores after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of frozen shoulder confirmed by an orthopedician.
* Patients in stage II or III of adhesive capsulitis.
* Participants of both genders aged 41-60 years.
* Subjects with a restricted range of motion (ROM), with losses of 25% or greater compared to the unaffected shoulder.

Exclusion Criteria:

* Rotator cuff tears.
* Overuse injuries.
* History of rheumatoid arthritis, osteoarthritis, or malignancies in the shoulder region.
* Adhesive capsulitis secondary to neurological disorders.
* Unstable shoulders or recurrent dislocations.
* Post-surgical cases involving the shoulder.

Ages: 41 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS | 12 Months
  Visual Analogue Scale (VAS) is one of the pain rating scales. Pain intensity can be categorized based on VAS scores, with mild pain typically ranging from 1-3, moderate pain from 4-6, and severe pain from 7-10.
Shoulder Pain and Disability Index (SPADI) | 12 Months
  The SPADI will be used to assess pain and disability. The pain subscale will measure the severity of pain during specific activities using a 0-10 numeric rating scale. The disability subscale will evaluate the difficulty experienced in performing daily activities involving the shoulder. SPADI scores will be recorded at the start of the treatment and again after completing the six treatment sessions to compare the changes in pain and functional status

CONTACTS AND LOCATIONS:
Locations (1):
- Gosha shifa hospital lahore gulshan ravi A block, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No